CLINICAL TRIAL: NCT04350853
Title: Surgical Extrusion for the Clinical Crown Lengthening: a 12-months Prospective Clinical Study
Brief Title: Surgical Extrusion for the Clinical Crown Lengthening: a 12-months Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Marc Llaquet Pujol, Principal investigator, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46150711
Record Dates: First submitted 2020-04-08; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Tooth Decay
Keywords: extrusion
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical extrusion group (Experimental): Surgical extrusion is performed in each patient of this group
  Interventions: Procedure: Surgical extrusion

INTERVENTIONS:
Procedure: Surgical extrusion — Surgically coronal reposition of the tooth

SUMMARY:
This is a prospective study in which surgical extrusion of single-rooted teeth is carried out by the same operator in 15 consecutive patients.

Main objective: to evaluate the soft tissue rebound of the teeth 1 year after the surgery.

Null hypothesis (H0): surgical extrusion is not a predictable treatment for the restoration of single rooted teeth.

ELIGIBILITY:
Inclusion Criteria:

* Systemically and periodontally healthy, non-smoking patients.
* Single-rooted, straight teeth with insufficient ferrule, which require restorative treatment.
* Teeth with a favorable crown-root ratio.

Exclusion Criteria:

* Severe systemic disease patients (American Society of Anesthesiologists classification 1 or 2).
* Multi-rooted, curved and/or short teeth.
* Teeth with an uncontrolled periodontal pathology.
* Pregnant women.
* Teeth with types ll or lll mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Soft tissue rebound | 12 months after the surgical extrusion
  mm
Tooth mobility (Miller classification) | 12 months after the surgical extrusion
  mm
Periapical lesion occurrence | 12 months after the surgical extrusion
  Assessed as the presence or not of a radiolucency at periapical radiograph (yes/no)
Patient's response to pain or discomfort at percussion test | 12 months after the surgical extrusion
  Patient's response measured by yes/no
Patient's response to pain or discomfort at palpation test | 12 months after the surgical extrusion
  Patient's response measured by yes/no
Root resorption occurrence | 12 months after the surgical extrusion
  Assessed as the presence or not of an inflammatory root resorption and a replacement root resorption at periapical radiograph

SECONDARY OUTCOMES:
Periodontal probing | 12 months after the surgical extrusion
  mm
Gum bleeding on periodontal probing (yes/no) | 12 months after the surgical extrusion
  Visual
Tooth plaque quantity | 12 months after the surgical extrusion
  Measured visually according to Turesky plaque index, in which the best score is 0 (no plaque) and the worst score is 5 (plaque covering 2/3 or more the crown of the tooth).
Interproximal papillae height | 12 months after the surgical extrusion
  Measured visually according to Jemt's index, in which the best score is 3 (interproximal space completely occupied) and the worst score is 0 (absent interproximal papilla).
Marginal bone loss | 12 months after the surgical extrusion
  mm
Crown-root ratio | 12 months after the surgical extrusion
  mm
Patient's satisfaction | 12 months after the surgical extrusion
  Measured visually using a visual analogue scale, in which the best score is 0 (highest level of patient's satisfaction) and the worst score is 10 (lowest level of patient's satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Marc Llaquet Pujol, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Collected data of the present study will be used for future research by the same research team.

REFERENCES:
- [Background] Kahnberg KE. Intra-alveolar transplantation. I. A 10-year follow-up of a method for surgical extrusion of root fractured teeth. Swed Dent J. 1996;20(5):165-72. PMID 9000325
- [Background] Kim SH, Tramontina V, Passanezi E. A new approach using the surgical extrusion procedure as an alternative for the reestablishment of biologic width. Int J Periodontics Restorative Dent. 2004 Feb;24(1):39-45. PMID 14984144
- [Background] Lee JH, Yoon SM. Surgical extrusion of multiple teeth with crown-root fractures: a case report with 18-months follow up. Dent Traumatol. 2015 Apr;31(2):150-5. doi: 10.1111/edt.12121. Epub 2014 Aug 11. PMID 25130861
- [Result] Elkhadem A, Mickan S, Richards D. Adverse events of surgical extrusion in treatment for crown-root and cervical root fractures: a systematic review of case series/reports. Dent Traumatol. 2014 Feb;30(1):1-14. doi: 10.1111/edt.12051. Epub 2013 Jun 25. PMID 23796195

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT04350853/Prot_SAP_ICF_000.pdf